CLINICAL TRIAL: NCT05962216
Title: Real-life Assessment of Brexpiprazole (Rexulti) in Schizophrenia and in Depressive Disorders: a Naturalistic Non-interventional Prospective Follow-up Study
Brief Title: Real-life Assessment of Brexpiprazole (Rexulti) in Schizophrenia and in Depressive Disorders
Acronym: ReSD
Status: Recruiting | Type: Observational
Sponsor: Dr. Albert Kar-Kin Chung (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Albert Kar-Kin Chung, Clinical Assistant Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Other Study IDs: ReSD-HK
Record Dates: First submitted 2023-07-03; First posted 2023-07-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Psychosis; Depression
MeSH Terms: conditions — Psychotic Disorders; Depression | interventions — brexpiprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole as treatment for psychosis and schizophrenia, and/or as augmentation treatment for depressive disorders
  Other Names: Rexulti

SUMMARY:
Not only being the mainstay of treatment for schizophrenia spectrum psychotic disorders, antipsychotics, especially the second-generation antipsychotics (SGAs) have also been recommended as augmenting agents for treating depression. Dopaminergic agents, including both dopamine D2/D3 antagonists and dopamine partial D2 agonists, have been effective for treating psychosis and schizophrenia. Amongst all SGAs, those with partial D2 agonistic property are generally acknowledged to have better side-effect profiles with lower incidence of extrapyramidal side-effects, prolactin increase, weight gain, QTc prolongation, and metabolic syndrome, as well as more efficacious in alleviating depressive symptoms. Up-to-date, three SGAs, namely aripiprazole, brexpiprazole and cariprazine, are known to possess such partial D2 agonism. ReSD-HK study is part of the ReSD Asian Study aiming to carefully evaluate a cohort of patients prescribed with brexpiprazole on its efficacy and tolerability as treatment for schizophrenia and/or depression in a real-life clinical setting.

DETAILED DESCRIPTION:
This is a 6-month, non-interventional, prospective naturalist study that adult patients (18-65 years old) receiving brexpiprazole for treatment of psychosis and/or as adjunctive treatment for major depressive disorder are eligible to participate. Minimal exclusion criteria are employed to fit the usual real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18- 65 years old at the time of enrollment
* Able to read and communicate in English and/or Chinese
* Able to give informed consent
* Has been diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5), or International Statistical Classification of Diseases and Related Health Problems 10th revision (ICD-10) to have either Psychotic Disorders (F10-F19.5, F20-23, F25, F32-F33)
* is receiving brexpiprazole as treatment for less than 4 weeks at the time of recruitment

Exclusion Criteria:

* Age <18 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Had been diagnosed to have Intellectual Disabilities (DSM-5) or Mental Retardation (ICD-10 F70-73)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from psychosis or depressive disorders who are treated with the oral medication, brexpiprazole
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Psychiatric Rating Scale-24 in 6 months | 6 months
  Efficacy measures the change from baseline, to that at 3rd and 6th months
Change in Clinical Global Impression in 6 months | 6 months
  Efficacy measures the change from baseline, to that at 3rd and 6th months
Change in Beck Anxiety Inventory in 6 months | 6 months
  Efficacy measures the change from baseline, to that at 3rd and 6th months
Change in Beck Depression Inventory in 6 months | 6 months
  Efficacy measures the change from baseline, to that at 3rd and 6th months
Change in Digital Symbol Substitution Test in 6 months | 6 months
  Efficacy measures the change from baseline, to that at 3rd and 6th months
Change in World Health Organization Disability Assessment Schedule 2.0 in 6 months | 6 months
  Efficacy measures the change from baseline, to that at 3rd and 6th months

SECONDARY OUTCOMES:
Glasgow Antipsychotic Side-effects Scale in 6 months | 6 months
  Tolerability measures at baseline, at 3rd and 6th months. Higher score means greater side-effects with the minimum score of 0 and the maximum score of 63.
Simpson-Angus Scale in 6 months | 6 months
  Tolerability measures at baseline, at 3rd and 6th months. The cut-off score is 3.
Barnes Akathisia Rating Scale in 6 months | 6 months
  Tolerability measures at baseline, at 3rd and 6th months. The cut-off score is 2.

OTHER OUTCOMES:
QTc interval | 6 months
  Tolerability measures at baseline and 6th months

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
To be shared within the ReSD Asian Study Group
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Five year after the study period upon the last subject recruitments in the respective study sites.
Access Criteria: For those named investigator who are engaged in the ReSD Asian Study with agreement signed.